CLINICAL TRIAL: NCT01134705
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 3 Clinical Study to Assess the Efficacy and Safety of BDP HFA Nasal Aerosol (320 Mcg, Once Daily) in the Treatment of Perennial Allergic Rhinitis (PAR) in Adult and Adolescent Subjects (12 Years of Age and Older)
Brief Title: Study in Adult and Adolescent Subjects With PAR (Perennial Allergic Rhinitis)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BDP-AR-302
Record Dates: First submitted 2010-05-27; First posted 2010-06-02 (Estimated); Results first posted 2012-05-23 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-04

CONDITIONS: Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BDP HFA 320 µg/day (Experimental): During the 6-week double-blind Treatment Period participants self-administered 4 actuations (two per nostril) of 80 µg BDP HFA once daily.
  Interventions: Drug: Beclomethasone dipropionate hydrofluoroalkane HFA Nasal Aerosol
- Placebo (Placebo Comparator): During the 6-week double-blind Treatment Period participants self-administered four actuations (two per nostril) of placebo HFA once daily.
  Interventions: Drug: Placebo Nasal Aerosol

INTERVENTIONS:
Drug: Beclomethasone dipropionate hydrofluoroalkane HFA Nasal Aerosol — Beclomethasone dipropionate (BDP) Hydrofluoroalkane (HFA) Nasal Aerosol
  Other Names: QNASL(TM)
  Arms: BDP HFA 320 µg/day
Drug: Placebo Nasal Aerosol — HFA Vehicle Aerosol
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the efficacy and safety of an investigational nasal aerosol compared with placebo nasal aerosol in the treatment of perennial allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Documented history of perennial allergic rhinitis
* A demonstrated sensitivity to at least one allergen known to induce PAR through a standard skin prick test.
* Minimum subject-reported reflective total nasal symptom score (rTNSS) of at least 6 (out of a possible 12)
* Other criteria apply

Exclusion Criteria:

* History of physical findings of nasal pathology (within 60 days prior to screening visit)
* Participation in any investigational drug study 30 days preceding screening visit
* History of respiratory infection/disorder with 14 days preceding screening visit or during the run-in period
* Use of any prohibited concomitant medications

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudeesh Tantry, Ph.D., Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (33):
- United States (33):
  - Teva Clinical Study Site, Los Angeles, California
  - Teva Clinical Study Site, Mission Viejo, California
  - Teva Clinical Study Site, San Diego, California
  - Teva Clinical Study Site, San Jose, California
  - Teva Clinical Study Site, Miami, Florida
  - Teva Clinical Study Site, Tallahassee, Florida
  - Teva Clinical Study Site, Lilburn, Georgia
  - Teva Clinical Study Site, Indianapolis, Indiana
  - Teva Clinical Study Site, Bangor, Maine
  - Teva Clinical Study Site, Bethesda, Maryland
  - Teva Clinical Study Site, Rolla, Missouri
  - Teva Clinical Study Site, St Louis, Missouri
  - Teva Clinical Study Site, Brick, New Jersey
  - Teva Clinical Study Site, Raleigh, North Carolina
  - Teva Clinical Study Site, Winston-Salem, North Carolina
  - Teva Clinical Study Site, Canton, Ohio
  - Teva Clinical Study Site, Medford, Oregon
  - Teva Clinical Study Site, Portland, Oregon
  - Teva Clinical Study Site, Blue Bell, Pennsylvania
  - Teva Clinical Study Site, Upland, Pennsylvania
  - Teva Clinical Study Site, Providence, Rhode Island
  - Teva Clinical Study Site, Charleston, South Carolina
  - Teva Clinical Study Site, Spartanburg, South Carolina
  - Teva Clinical Study Site, Austin, Texas
  - Teva Clinical Study Site, Dallas, Texas
  - Teva Clinical Study Site, Fort Worth, Texas
  - Teva Clinical Study Site, Katy, Texas
  - Teva Clinical Study Site, New Braunfels, Texas
  - Teva Clinical Study Site, San Antonio, Texas
  - Teva Clinical Study Site, Waco, Texas
  - Teva Clinical Study Site, Newport News, Virginia
  - Teva Clinical Study Site, Richmond, Virginia
  - Teva Clinical Study Site, Bellevue, Washington

REFERENCES:
- [Result] Meltzer EO, Jacobs RL, LaForce CF, Dorinsky PM, Kelley L, Dunbar SA, Tantry SK (2011). BDP HFA Nasal Aerosol 320 µg Once Daily Is Safe and Effective in the Treatment of Nasal Symptoms Associated With Perennial Allergic Rhinitis. Ann Allergy Asthma Immunol. 107(11):A118.
- [Result] Meltzer EO, Jacobs RL, LaForce CF, Dorinsky PM, Kelley L, Dunbar SA, Tantry SK. . BDP HFA Nasal Aerosol 320 µg Once Daily Is Safe and Effective in the Treatment of Nasal Symptoms Associated With Perennial Allergic Rhinitis. Ann Allergy Asthma Immunol (Supplement); 107(11):A118 - Poster presentation.
- [Result] Carr W, Meltzer EO, Finn A, Dorinsky PM, Kelley L, Dunbar SA, Tantry SK. Effective nasal symptom relief and improvement in health-related quality of life in subjects with perennial allergic rhinitis following 6-week
- [Derived] Meltzer EO, Korenblat PE, Lanier BQ, Kelley L, Tantry SK. Beclomethasone dipropionate nasal aerosol with an integrated dose counter: functionality and performance. Allergy Asthma Proc. 2013 Nov-Dec;34(6):534-41. doi: 10.2500/aap.2013.34.3707. PMID 24169062
- [Derived] Nayak AS, Atiee GJ, Dige E, Maloney J, Nolte H. Safety of ragweed sublingual allergy immunotherapy tablets in adults with allergic rhinoconjunctivitis. Allergy Asthma Proc. 2012 Sep-Oct;33(5):404-10. doi: 10.2500/aap.2012.33.3605. PMID 23026182
- [Derived] Meltzer EO, Jacobs RL, LaForce CF, Kelley CL, Dunbar SA, Tantry SK. Safety and efficacy of once-daily treatment with beclomethasone dipropionate nasal aerosol in subjects with perennial allergic rhinitis. Allergy Asthma Proc. 2012 May-Jun;33(3):249-57. doi: 10.2500/aap.2012.33.3571. PMID 22737708

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 675 patients were screened and 574 patients were enrolled in the study and participated in the Run-in Period. Of the 574 enrolled patients, 474 were randomized to study treatment.
Pre-assignment Details: During the 7 to 21 day Run-in Period, participants self-administered a single-blind placebo nasal aerosol once daily in the morning and assessed and recorded their twice daily allergic rhinitis symptoms to determine eligibility for randomization.
Groups:
- BDP HFA 320 µg/Day: During the 6-week double-blind Treatment Period participants self-administered 4 actuations (two per nostril) of 80 micrograms (µg) beclomethasone dipropionate (BDP) hydrofluoroalkane (HFA) once daily.
Period: Overall Study
Arm/Group | BDP HFA 320 µg/Day | Placebo
Started | 236 | 238
Intent to Treat Population | 232 (Participants who received at least 1 dose of study drug and had at least 1 post-baseline assessment.) | 234 (Participants who received at least 1 dose of study drug and had at least 1 post-baseline assessment.)
Completed | 221 | 216
Not Completed | 15 | 22
Not completed — Adverse Event | 1 | 7
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Pregnancy | 1 | 0
Not completed — Lost to Follow-up | 5 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Other | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BDP HFA 320 µg/Day | Placebo | Total
Number analyzed (Participants) | 232 | 234 | 466
Age Continuous [Mean (Standard Deviation); unit: years] — Demographic data are provided for the Intent to Treat population.
  years | 36.8 (14.5) | 37.2 (13.7) | 37.0 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 161 | 319
  Male | 74 | 73 | 147
Race/Ethnicity, Customized [Number; unit: participants] — A participant may select more than one race type.
  participants
    White | 186 | 185 | 371
    Black or African American | 40 | 40 | 80
    Asian | 6 | 5 | 11
    American Indian or Alaskan Native | 1 | 2 | 3
    Other | 1 | 6 | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 26 | 30 | 56
  Not Hispanic or Latino | 206 | 204 | 410
Region of Enrollment [Number; unit: participants]
  United States | 232 | 234 | 466

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average AM and PM Reflective Total Nasal Symptom Score (rTNSS) Over the Six-week Treatment Period
Description: Participants recorded the severity of their nasal symptoms (sneezing, runny nose, itchy nose and nasal congestion) over the past 12 hours twice daily (AM & PM) using the following scale:
  0=absent (no sign/symptom); 1=mild (sign/symptom present, awareness, easily tolerated); 2=moderate (awareness of sign/symptom, bothersome but tolerable); 3=severe (sign/symptoms hard to tolerate, interfere with daily activities and/or sleeping).
  The total nasal symptom score (sum of 4 symptom scores) ranges from 0 to 12 (worst symptoms). A negative change from Baseline score indicates symptom improvement.
Time Frame: Baseline (Days -3 to 0) and Days 1-43 (6-week Treatment Period)
Population: Intent-to-Treat (ITT) Population: The ITT population included all randomized patients who received at least one dose of randomized study medication and had at least one post-baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 232 | 234
units on a scale | -2.5 (0.14) | -1.6 (0.14)
Statistical Analysis 1: Comparison: BDP HFA 320 µg/Day vs Placebo; Test type: Superiority or Other; p < 0.001, Repeated measures Analysis of covariance — A priori threshold for statistical significance is p<0.05; The repeated measures ANCOVA included covariate adjustment for baseline, day, treatment, and the treatment by day interaction; LS Mean Difference = -0.84, 95% CI 2-sided [-1.2 to -0.5]

2. Secondary Outcome: Change From Baseline in Average AM and PM Instantaneous Total Nasal Symptom Score (iTNSS) Over the Six-week Treatment Period
Description: Participants recorded the severity of their nasal symptoms (sneezing, runny nose, itchy nose and nasal congestion) over the 10 minutes prior to assessment twice daily (AM & PM) using the following scale:
  0=absent (no sign/symptom); 1=mild (sign/symptom present, easily tolerated); 2=moderate (awareness of symptoms, bothersome but tolerable); 3=severe (symptoms hard to tolerate, interfere with daily activities and/or sleeping).
  The total nasal symptom score (sum of the 4 symptom scores) ranges from 0 to 12 (worst symptoms). A negative change from Baseline score indicates symptom improvement.
Time Frame: Baseline (Days -3 to 0) and Days 1-43 (6-week Treatment Period)
Population: Intent to treat population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 232 | 234
units on a scale | -2.1 (0.13) | -1.4 (0.13)
Statistical Analysis 1: Comparison: BDP HFA 320 µg/Day vs Placebo; Test type: Superiority or Other; p < 0.001, Repeated measures ANCOVA — A priori threshold for statistical significance is p<0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.78, 95% CI 2-sided [-1.1 to -0.4]

3. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ)
Description: The adult RQLQ has 28 questions in 7 domains (activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms, and emotional). Participants were asked to recall their experiences during the previous week and to give their responses on a 7-point scale (0 = Least severe to 6 = Extremely severe). The overall RQLQ score is the mean of all 28 responses, and ranges from 0 to 7. A negative change from Baseline score indicates improvement.
Time Frame: Baseline and Week 6
Population: The RQLQ population included adults (18 years and older) with an impaired quality of life at Baseline as defined by a RQLQ score at the Randomization Visit of 3.0 or greater.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 132 | 125
units on a scale | -1.5 (0.14) | -0.9 (0.14)
Statistical Analysis 1: Comparison: BDP HFA 320 µg/Day vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA — A priori threshold for statistical significance is p<0.05; ANCOVA with treatment, baseline and center in the model; LS Mean Difference = -0.58, 95% CI 2-sided [-0.9 to -0.2]

ADVERSE EVENTS:
Arm/Group | BDP HFA 320 µg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 1/236 | 0/238
Other Adverse Events (participants affected / at risk) | 14/236 | 12/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BDP HFA 320 µg/Day (N=236) | Placebo (N=238)
Arrhythmia (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BDP HFA 320 µg/Day (N=236) | Placebo (N=238)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 14 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.